CLINICAL TRIAL: NCT04447625
Title: Introducing Intrauterine Antibiotic Infusion as a Novel Approach in Effectively Treating Chronic Endometritis and Restoring Reproductive Dynamics: A Pilot Study
Brief Title: Intrauterine Antibiotic Infusion in Treating Chronic Endometritis and Restoring Reproductive Dynamics
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genesis Athens Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1A
Record Dates: First submitted 2020-06-20; First posted 2020-06-25 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Chronic Endometritis
Keywords: CE treatment; infertility; oral antibiotic administration; intrauterine antibiotic infusion
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CE patients receiving OAA (Active Comparator): Patients diagnosed with CE receiving the gold standard treatment of oral antibiotic administration (OAA)
  Interventions: Drug: Oral antibiotic administration
- CE patients receiving OAA and IAI (Experimental): Patients diagnosed with CE receiving a combination of the gold standard treatment of oral antibiotic administration (OAA) and intrauterine antibiotic infusion (IAI)
  Interventions: Drug: Oral antibiotic administration; Drug: Intrauterine antibiotic infusion

INTERVENTIONS:
Drug: Oral antibiotic administration — per os antibiotic administration as the standard line of strategy for treating CE of doxycycline at a dosage of 100mg twice a day for 14 days and metronidazole of 500mg twice a day for 14 days
Drug: Intrauterine antibiotic infusion — intrauterine infusion of 3ml of ciprofloxacin at a concentration of 200 mg/100 ml
  Arms: CE patients receiving OAA and IAI

SUMMARY:
Chronic Endometritis (CE) is related to infertility and entails a challenging management. This study investigates the treatment of off-label intrauterine antibiotic infusion (IAI) combined with oral antibiotic administration (OAA), and it assesses respective performance against the gold standard treatment of OAA. Data sourced herein reports on treatment efficiency and fertility restoration for both patients aiming to conceive naturally or via In Vitro fertilization (IVF).

ELIGIBILITY:
Inclusion Criteria:

* Positive diagnosis of CE
* Recurrent Pregnancy Loss (RPL) or Recurrent Implantation Failure (RIF)
* No previous live birth
* FSH and LH levels -evaluated on day 2 of the menstrual cycle- <12 IU/ml
* AMH levels >1.1ng/ml
* Progesterone levels -evaluated on day 21 of the menstrual cycle- > 2 and <25 ng/ml
* 18.5<BMI<29.9
* 18<Patients' age<40

Exclusion Criteria:

* Diagnosed endometriosis or other related Pelvic Inflammatory Disorder (PID)
* Current or previous cancer diagnosis
* Auto-immune, genetic or reproductive disorders
* Reproductive history of pregnancy loss due to genetic abnormalities
* Male factor infertility diagnosis

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2020-01-03 (Actual)

PRIMARY OUTCOMES:
Treatment efficiency rate | Treatment efficiency rate was assessed immediately after treatment completion
  Negative results in all three diagnostic evaluations of CE namely hysteroscopic investigation, endometrial biopsy, along with histological analysis and microbiological culture indicating successful treatment of CE
Side-effects rate | Side-effects were monitored from treatment initiation until completion of treatment. Treatment duration: 14 days for Arm 1 and 30 days for Arm 2
  Number of reports of minimal, mild, and moderate side-effects per treated patients

SECONDARY OUTCOMES:
Clinical pregnancy rate | Clinical pregnancy rate was assessed 6-7 weeks following last menstrual period for patients that achieved a pregnancy. A time frame of 6 months was allowed for patients to achieve a pregnancy post treatment.
  Clinical pregnancy rate was defined by the presence of a fetal heartbeat at 6-7 weeks following last menstrual period (LMP)
Live birth rate | A time frame of 40-41 weeks was allowed to assess live birth rate following patients' last menstrual period.
  Number of live births per clinical pregnancy

CONTACTS AND LOCATIONS:
Locations (1):
- Human Reproduction LTD, Athens, Holargos, Greece

IPD SHARING:
Plan to Share IPD: No